CLINICAL TRIAL: NCT03465397
Title: Multicenter, Randomized Study to Evaluate the Effectiveness of the Individualization of the Immunological Risk Based on Biomarkers (Disparity of HLA and IFN-γ ELISPOT) to Optimize Immunosuppressor Treatment in Living-donor Renal Recipients
Brief Title: Individualization of the Immunological Risk Based on Selective Biomarkers in Living-donor Renal Recipients
Acronym: BIOIMMUN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ORIOL BESTARD (Other)
Collaborators: Department of Health, Generalitat de Catalunya (Other Government)
Responsible Party: Sponsor-Investigator, ORIOL BESTARD, Head of Transplant Unit, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BIOIMMUN
Record Dates: First submitted 2018-01-04; First posted 2018-03-14 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Kidney Transplant Failure and Rejection
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Intervention Model Description: Multicenter open clinical trial, randomized, stratified by age, parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental (Experimental): Biomarkers driven immunosuppressive therapy: the immunosuppressive treatment of the patients is determined according to the result of 2 biomarkers of immunological risk
  Interventions: Diagnostic Test: biomarkers driven immunosuppressive therapy
- control (No Intervention): All patients receive the usual triple immunosuppressive treatment, without depending on the results of any biomarker.

INTERVENTIONS:
Diagnostic Test: biomarkers driven immunosuppressive therapy — the immunosuppressive treatment of the patients is determined according to the result of 2 biomarkers of immunological risk
  Arms: experimental

SUMMARY:
This is a clinical trial comparing the immunosuppressive treatment determined according to two biomarkers, donor-specific IFN-γ ELISPOT and Mismatch of HLA between donor and recipient, in patients undergoing low immunological risk live donor kidney transplantation

DETAILED DESCRIPTION:
This is a national multicenter clinical trial, controlled, randomized, stratified, parallel groups, and without masking.

This is a prospective intervention study in which two strategies for determining immunosuppressive treatment in kidney transplant patients from a live donor with low immunological risk are compared according to solid phase antibody detection techniques (cPRA 0% and isolated negative antigen) and crossmatch by negative cytotoxicity. Patients are randomized in a 1: 1 ratio to receive one of two immunosuppressive treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women (≥18 years).
2. Receptors of a first kidney transplant from an incompatible HLA living donor (at least 1 mismatch HLA at any antigenic level).
3. AB0 compatible transplant.
4. Patients with a calculated PRA of 0% by solid phase technique and absence of anti-HLA class I and class II antibodies by single antigen test (Luminex®).
5. Patients who agree to participate in the Trial by signing the Specific Informed Consent of this study.
6. Potentially fertile women should use high reliability contraceptive methods (Pearl-Index <1) in order to avoid pregnancy during the entire duration of the study and up to 6 weeks after the end of their treatment with Mycophenolate Mofetil (MMF). Potentially Fertile Women include any woman who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or who is not post-menopausal (defined as amenorrhea ≥ 12 consecutive months, or women who are receiving hormone replacement therapy with a documented level of follicle stimulating hormone (FSH)> 35 mlU / ml). Potentially fertile women must have a pregnancy test with a negative result in the 72 hours prior to the start of the trial.
7. Sexually active males (including vasectomized males) who are being treated with MMF must accept the use of barrier contraceptive methods during MMF treatment and for 90 days thereafter. Potentially fertile partners of these patients should use a reliable contraceptive method during the same period, in order to minimize the risk of pregnancy.
8. Patients must agree not to donate blood during treatment with MMF and during the 6 subsequent weeks. Males should not make a sperm donation during MMF treatment and up to 90 days after completion.

Exclusion Criteria:

1. Patients with a calculated PRA higher than 0% per solid phase and / or anti-HLA class I and / or class II antibodies detectable by single antigen test (Luminex®).
2. Positive result of Cross Match.
3. Patients who receive a graft from a cadaver donor.
4. Identical HLA patients
5. Patients who have undergone a previous solid organ transplant (including kidney transplant) or who are going to receive another solid organ transplant concomitantly.
6. Patients with any of the following basic renal diseases:

   * Glomerular primary focal and segmental sclerosis
   * Atypical hemolytic uremic syndrome (aHUS) / thrombotic thrombocytopenic purpura syndrome.
7. Patients with chronic infection with Hepatitis B virus (HBV) and / or active infection with Hepatitis C virus (positive PCR result) at the time of transplant.
8. Patients with infection with the known Human Immunodeficiency Virus (HIV).
9. Patients with active systemic infection that requires the continued administration of antibiotics.
10. Patients with any neoplasm except localized skin cancer and who is receiving adequate treatment.
11. Patients with severe anemia (hemoglobin <6g / dl), leukopenia (WBC <2500 / mm3) and / or thrombocytopenia (platelets <80,000 / mm3).
12. Patients who are hemodynamically unstable even if they have hemoglobin levels> 6g / dL.
13. Patients with intestinal pathology or severe diarrhea that may decrease absorption according to medical criteria.
14. Patients with known hypersensitivity to any of the drugs used in this study.
15. Patients who have received any investigational drug in the 30 days prior to their inclusion in this study.
16. Potentially fertile women who do not agree to use reliable contraceptive measures during the trial, who are pregnant, breastfeeding or who present a positive pregnancy test at the time of their inclusion in the study.
17. Patients who are legally detained in an official institution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2017-11-10 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
composite | 24 months
  composite variable evaluated at 2 years of follow-up as a proportion of patients who meet any of the following criteria: loss of renal function, incidence of acute clinical rejection confirmed by biopsy (BPAR) and development of dnDSA.

SECONDARY OUTCOMES:
mortality | 24 months
  Mortality from any cause
kidney graft loss | 24 months
  Loss of kidney graft
Subclinical and chronic rejection | at 3 and 24 months
  Incidence and severity of subclinical and chronic rejection (according to protocol biopsies)
Opportunistic infections | 24 months
  Incidence of opportunistic infections
Metabolopathies | 24 months
  Incidence of metabolopathies derived from the treatment (diabetes mellitus, dyslipidemia and HT)
Cardiovascular Events | 24 months
  Incidence of cardiovascular events
Malignancy | 24 months
  Incidence of malignancy (cutaneous and non-cutaneous cancer)
Treatment maintenance | 24 months
  Proportion of patients who maintain the treatment according to the protocol at the end of the trial.
Immune Response Changes | 24 months
  Changes in the immune response at 24 months according to the biomarkers (urine cytokines CXCL9 and CXCL10, test KSORT, ELISPOT)
Economic cost | 24 months
  Study of the economic cost
Serious adverse reactions | 24 months
  serious adverse events with a possible causal relationship with the immunosuppressive treatment)

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Germans Trias I Pujol, Badalona
  - Fundació Puigvert, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital Del Mar, Barcelona
  - Hospital Universitari Vall D'Hebrón, Barcelona